CLINICAL TRIAL: NCT06012942
Title: Prevalence and Long Term Effects of Frailty in Elderly Intensive Care Patients
Acronym: SkrInt
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital of North Norway (Other)
Collaborators: The Royal Norwegian Ministry of Health (Other); Haukeland University Hospital (Other); University Hospital, Akershus (Other); Trondheim University Hospital (Other); Bodø Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: HNF1632-22
Record Dates: First submitted 2023-02-22; First posted 2023-08-28 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-02

CONDITIONS: Frailty; Critical Illness
Keywords: clinical frailty scale; mechanical ventilation; elderly; EQ-5D-5L
MeSH Terms: conditions — Frailty; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary aim is to study change of critical frailty scale (CFS) and health related quality of life (EQ-5D-5L) in a long-term follow-up of ICU survivors. We aim to identify important ICU related predictors for change in CFS and EQ-5D-5L in long term follow up (1 yr).

Secondary aim is to investigate how CFS pre-admission is related to intrahospital treatment intensity level, severity score and mortality.

DETAILED DESCRIPTION:
This is a multi-centre norwegian observational, prospective multicenter Norway coordinated from University hospital North Norway, Tromso.

The study is approved by The Regional Committee for Medical Research Ethics Northern Norway.

The following scores will be assessed by asking the patient and relative during ICU stay: CFS, EQ5DL before current critical illness.

The following demographic and clinical data will be retrieved from the medical records: Comorbidity before critical illness, reasons for ICU admission, daily severity score (SOFA- score), length of mechanical ventilation, dialysis, tracheostomy, Habitat before and after ICU treatment, ICU and hospital length of stay, complications retrieved during intensive care treatment, mortality, limitation of treatment.

The patients will be followed up with telephone interview after hospital discharge for evaluation of: Comorbidity, CFS, EQ5DData for all sites are collected and managed using RedCap electronic data capture tools.

Three research nurses will do the follow up with telephone interviews on all sites and record the data in RedCap.

We aim to enroll 300 patients before 31. Des 2024.

ELIGIBILITY:
Inclusion Criteria:

* >= 65 years
* ≥ 24 hours mechanical ventilation
* Written informed consent from patient or next of kin

Exclusion Criteria:

* Readmission of patient included in the study
* Not possible to obtain a valid CFS or and EQ-5D-5L at admission or follow-up of CFS because of social context or language.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: ICU patients above 65 years old requiring invasive mechanical ventilation> 24 hours are screened for inclusion during the intensive care stay.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-07-07 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Clinical frailty score | Change in Clinical Frailty score from 3 months to 12 months follow up
  Score from 1 to 9.
EuroQol 5-Dimension 5-Level (EQ-5D-5L) | Change in EQ-5D-5L from 3 months to 12 months
  The scale measures quality of life on a 5-component scale
Mortality | ICU-stay or subsequent 12 months.
  Mortality during ICU-stay or subsequent 12 months.

SECONDARY OUTCOMES:
ICU readmission | Long-term follow up (1 yr)
  ICU readmission rate
ICU-LOS | Through total ICU stay, up to 3 months
  ICU length of stay
Treatment intensity level | From inclusion in the study to discharge from intensive care unit, up to three months.
  ICU treatment intensity level

CONTACTS AND LOCATIONS:
Overall Officials: Shirin K Frisvold, MD/PhD, Principal Investigator — University Hospital of North Norway
Locations (5):
- Norway (5):
  - Akershus University hospital, General Intensive care department, Lørenskog, Nordbyhagen
  - Haukeland University hospital, General Intensive care unit, Bergen
  - Nordlandssykehuset Bodø, Intensivavdelingen, Bodø
  - University Hospital of North Norway, Tromsø
  - Trondheim University hospital, General Intensive care department, Trondheim

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported, after deidentification (text, tables, figures and appendices).
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 12 months and ending 5 years following article publication.
Access Criteria: The presented dataset will be considered available from the corresponding author on reasonable request based on formal national approvals.

REFERENCES:
- [Background] Flaatten H, De Lange DW, Morandi A, Andersen FH, Artigas A, Bertolini G, Boumendil A, Cecconi M, Christensen S, Faraldi L, Fjolner J, Jung C, Marsh B, Moreno R, Oeyen S, Ohman CA, Pinto BB, Soliman IW, Szczeklik W, Valentin A, Watson X, Zaferidis T, Guidet B; VIP1 study group. The impact of frailty on ICU and 30-day mortality and the level of care in very elderly patients (>/= 80 years). Intensive Care Med. 2017 Dec;43(12):1820-1828. doi: 10.1007/s00134-017-4940-8. Epub 2017 Sep 21. PMID 28936626
- [Background] Flaatten H, Beil M, Guidet B. Prognostication in older ICU patients: mission impossible? Br J Anaesth. 2020 Nov;125(5):655-657. doi: 10.1016/j.bja.2020.08.005. Epub 2020 Aug 14. No abstract available. PMID 32868042
- [Derived] Kroken BA, Bergum D, Berg KS, Espinasse M, Fossum OK, Garratt AM, Klepstad P, Kvale R, Strand B, Flaatten HK, Frisvold SK. Frailty and health-related life quality in long-term follow up of intensive care patients above 65 years old: Protocol for a Norwegian prospective, observational multicenter study. Acta Anaesthesiol Scand. 2024 Nov;68(10):1595-1600. doi: 10.1111/aas.14532. Epub 2024 Oct 1. PMID 39353584